CLINICAL TRIAL: NCT06097611
Title: Efficacy and Outcome of Early Administration of Tranexamic Acid in Pediatric Polytraumatized Patients
Brief Title: Tranexamic Acid Effect in Pediatric
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaaban Hassan Hassan Salim, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Tranexamic Acid Effect
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Tranexamic Acid Effect in Pediatric Polytraumatized Patients
Keywords: Tranexamic Acid; Effect; Polytrauma; Pediatric
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Efficacy of early Tranexamic Acid in Pediatric Polytraumatized Patients (Experimental)
  Interventions: Drug: Tranexamic Acid administration
- Efficacy of Early Tranexamic Acid in Pediatric Polytraumatized Patients (Active Comparator)
  Interventions: Drug: Tranexamic Acid administration

INTERVENTIONS:
Drug: Tranexamic Acid administration — Tranexamic Acid administration to compare mortality and blood transfusion amounts among severely polytraumatized pediatrics who did or did not receive tranexamic acid within 3 h of injury

SUMMARY:
The study will compare mortality and blood transfusion amounts among severely polytraumatized pediatrics who did or did not receive tranexamic acid within 3 h of injury, based on Injury Severity Score (ISS) and indicators of coagulopathy and fibrinolysis.

DETAILED DESCRIPTION:
Trauma is a leading cause of mortality in the pediatric population. In 2008, the American Academy of Pediatrics noted that trauma accounts for more deaths than all other causes combined . Bleeding remains the most preventable cause of death after trauma. A major recent advance was the recognition that coagulation defects are greatly responsible for the disproportional mortality caused by bleeding. Managing coagulation defects has become a forefront issue in trauma and novel strategies proposed include hemostatic resuscitation, adoption of massive transfusion protocols and other innovations , most with little evidence to support them. The exception is the proposal to administer tranexamic acid (TXA) to bleeding adult trauma patients.

To date, no medical treatment has been shown to reduce mortality in the setting of pediatric trauma; however, this evidence does exist in adults. Bleeding and coagulopathy due to trauma are associated with mortality in both adults and children. Clinical research has demonstrated a reduction in trauma-related mortality with early use of TXA in adult patients in both civilian and military settings . In adult patients with hemodynamic instability and ongoing bleeding, TXA is expected to save 1 in 67 lives . There is no scientific or biological reason to suggest that a similar mortality benefit will not be seen in pediatric trauma. The investigators feel the incorporation of TXA into pediatric trauma management has the potential to also significantly reduce mortality in children and youths, without increasing adverse events. This review explores the hematologic differences and similarities between injured children and adults, and the idea that TXA may be a novel and promising treatment in pediatric hemorrhagic trauma despite the current lack of evidence for its use in this setting.

TXA is an antifibrinolytic that reversibly binds to plasminogen at the lysine binding site, thus preventing the binding of plasmin (ogen) to fibrin and the subsequent degradation of fibrin . It is a generic, inexpensive medication used to prevent fibrin breakdown and reduce bleeding in various clinical settings (including orthopedic and cardiovascular surgery, post-partum hemorrhage, gastrointestinal hemorrhage, epistaxis, certain ophthalmologic conditions and other obstetric/gynecologic emergencies)

ELIGIBILITY:
Inclusion Criteria:

1. ISS ≥ 16
2. age 2-18 years
3. both genders
4. polytraum a

Exclusion Criteria:

1. age < 2 OR >18 years
2. period from injury to admission >6 hours
3. ISS<16
4. comorbidity with bleeding disorder, malignancy.
5. Patients receiving anticoagulant drugs.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Determine the mortality rate among polytraumatic pediatrics who received Tranexamic acid within 3 hours versus those who did not received | 1 yaer